CLINICAL TRIAL: NCT06716463
Title: PREdicting Failure of Non-inVasIve Ventilatory Support Using Non-invaSIve mONitoring in Non-intubated Patients With Acute Hypoxemic Respiratory Failure or Post-extubation Failure: the PREVISION Study
Brief Title: PREdicting Failure of Non-inVasIve Ventilatory Support Using Non-invaSIve mONitoring in Non-intubated Patients With Acute Hypoxemic Respiratory Failure or Post-extubation Failure. The PREVISION Study
Acronym: PREVISION
Status: Recruiting | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: Unity Health Toronto
Record Dates: First submitted 2024-11-25; First posted 2024-12-04 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Ventilatory Failure; Hypoxemic Respiratory Failure; Weaning Failure; Respiratory
Keywords: Electrical impedance tomography; High flow nasal cannula; Non-invasive ventilation; Diaphragm; Weaning failure; Post-extubation; Hypoxemic respiratory failure
MeSH Terms: conditions — Hypoventilation; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to assess the potential non-invasive tools (e.g. regional ventilation, respiratory muscle response, lung mechanic's parameters) to identify the risk of failure when using high flow nasal cannula (HFNC) or non-invasive ventilation (NIV).

The main question, it aims to answer is:

Does abnormal regional ventilation could predict HFNC or NIV failure?

DETAILED DESCRIPTION:
This is a single-center, prospective, physiological study.

The study will enroll patient who has used either HFNC or NIV for the indications of 1. to prevent worsening acute hypoxemic respiratory failure or 2. to prevent reintubation. Once being confirmed to meet the inclusion criteria, the research team will apply the electrical impedance tomography (EIT) on the patient and start recording for 5-10 minutes as well as perform diaphragm and parasternal intercostal muscle ultrasound when the patient is using HFNC or NIV. The current HFNC or NIV setting, some lung mechanic's parameters (e.g. rapid shallow breathing trial (RSBI), negative airway pressure generated during the first 100 milisecond (P0.1), end-expiratory occlusion pressure(ΔPocc) derived from NIV machine), patient's characteristic, dyspnea scores (intensive care respiratory distress observation scale, IC-RDOS; work of breathing scale; self-report of dyspnea visual analog scale, D-VAS), ICU and hospital length of stay will be also collected.

The investigator will use EIT to visualize where air goes in the patient's lung and inspiratory muscle ultrasonography (diaphragm and parasternal intercostal muscle) to visualize the muscle activities when using HFNC or NIV. EIT is a measurement often used in the ICU since it allows easy visualization and is a non-invasive technique. The sensors measure electrical current changes during inspiration and expiration and will not cause any pain or radiation concerns. The EIT belt (3-cm diameter) will be placed around the chest without causing adverse event/discomfort/pain.

The duration of study will be approximately 30 minutes. The study will be conducted one time for one enrolled patient.

HFNC or NIV (device) failure is considered as either intubation/reintubation or death, whatever has come first. It will be followed up to 7 days.

The investigators will proceed with the measurements only with agreement from the clinical team. The investigators will analyze the data collected offline with a dedicated software afterwards.

After these study procedures are completed, data will also be collected from the participant's chart and combined with relevant information from the HFNC or NIV settings and vital functions. Confidentiality will be maintained throughout the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Age of ≥ 18 years
* Using NIV or HFNC anywhere in the hospital

Exclusion Criteria:

* Chronic CO2 retention
* Neuromuscular disorder
* Requiring home NIV (CPAP or BIPAP)
* Tracheostomy
* Contraindication to EIT placement: pacemaker/defibrillator implantation, burns at the area of EIT placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who is using high flow nasal cannula (HFNC) or non-invasive ventilation (NIV) to either prevent 1. intubation in the context of acute hypoxemic respiratory failure or 2. reintubation in the context of high risk group of extubation.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Difference in regional ventilation distribution (%) | The parameter is measured at the time of enrolment. Failure of HFNC or NIV is adjudicated at 7 days.
  The primary endpoint is to assess regional ventilation distribution (%) when using HFNC or NIV to predict a device failure.

SECONDARY OUTCOMES:
Diaphragm or parasternal intercostal muscle thickening fraction | The parameter is measured at the time of enrolment. Failure of HFNC or NIV is adjudicated at 7 days.
  To assess ultrasound measurement of inspiratory muscle activity when using HFNC or NIV to predict a device failure.
Rapid shallow breathing index (RSBI) in mL/breaths/min | The parameter is measured at the time of enrolment. Failure of HFNC or NIV is adjudicated at 7 days.
  To assess non-invasive respiratory - rapid shallow breathing index (RSBI) derived from NIV to predict a device failure.
Respiratory drive using negative airway pressure generated during the first 100 millisecond (P0.1) | The parameter is measured at the time of enrolment. Failure of HFNC or NIV is adjudicated at 7 days.
  To assess respiratory drive - using negative airway pressure generated during the first 100 millisecond (P0.1) in cmH2O to predict device failure.
Respiratory effort using end-expiratory airway occlusion pressure (ΔPocc) | The parameter is measured at the time of enrolment. Failure of HFNC or NIV is adjudicated at 7 days.
  To assess respiratory effort using end-expiratory airway occlusion pressure (ΔPocc) in cmH2O to predict device failure
The intensive care respiratory distress observation scale (IC-RDOS) | The parameter is measured at the time of enrolment. Failure of HFNC or NIV is adjudicated at 7 days.
  To assess the level of dyspnea using intensive care respiratory distress observation scale (IC-RDOS) to predict a device failure. There is no minimum or maximum range depending on patient's heart rate, the higher score means worse outcome. When the score ≥ 2.4, it likely indicates clinically important dyspnea requiring clinical management.
The work of breathing scale | The parameter is measured at the time of enrolment. Failure of HFNC or NIV is adjudicated at 7 days.
  To assess the work of breathing scale to predict a device failure. Minimum is 3 and maximum is 12, the higher score means worse outcome. When the score > 4, it likely indicates severe respiratory distress.
Self-report of dyspnea visual analog scale (D-VAS) | The parameter is measured at the time of enrolment. Failure of HFNC or NIV is adjudicated at 7 days.
  To assess self-report of dyspnea visual analog scale (D-VAS) to predict a device failure. Minimum is 0 and maximum is 10, the higher score means worse outcome. When the score > 3, it likely indicates dyspnea and being used for quality of palliative care unit

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No